CLINICAL TRIAL: NCT05784285
Title: BEYOND: Body-function Enhancement for YOuth Through participatioN in Real-worlD Contexts. The Downstream Effects of Personalized 'Top-down' Participation-based Interventions Among Youth With Physical Disabilities
Brief Title: Downstream Effects of Personalized 'Top-down' Participation-based Interventions Among Youth With Physical Disabilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other); Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 480889
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries; Spina Bifida; Musculoskeletal Disorder; Juvenile Arthritis; Amputation; Cerebral Palsy
Keywords: participation; environmental barriers; youth; disabilities; body functions
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Dysraphism; Musculoskeletal Diseases; Arthritis, Juvenile; Cerebral Palsy | interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: A 22-week interrupted time series design with multiple baselines across 150 youth with physical disabilities stratified by sex and severity will be employed.
Masking Description: All assessors will be blinded to the time point in which the intervention begins and to the chosen activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based activity program (Experimental): Engagement in 8-week community-based activity program.
  Interventions: Behavioral: Engagement in a 8-week community-based activity program

INTERVENTIONS:
Behavioral: Engagement in a 8-week community-based activity program — Participants engage in a 8-week community-based activity program of their choice. In order to engage in the selected activity, an Occupational Therapist (OT) will meet with each youth in their home. Using the PREP 5 steps (Make goals; Map out a plan; Make it happen; Measure the process and outcomes; Move forward) the youth will choose a community program. The OT will then search for the appropriate program, identify and remove potential environmental barriers for participation in that activity (e.g., accessibility, equipment) and educate program instructors regarding the youth's specific needs. This process, which includes up to 12 hours of working with the OT, will set the stage for enrolment of the youth in a community program for a period of 8 weeks - the actual intervention phase.
  Other Names: Pathways and Resources for Engagement and Participation (PREP)

SUMMARY:
Participation in community-based activities is essential to the health and well-being of youth with physical disabilities; yet, it is extremely restricted. Emerging treatment approaches aimed at improving participation have shifted from focusing only on impaired body functions towards the performance of functional meaningful activities within the youth's natural environment. Investigators' initial results from studies in Quebec show that targeting intervention at the activity/participation level can result in improvement of impaired body functions (e.g., balance, attention, anxiety) - important components to address in rehabilitation. Investigators' team aims to continue studying the impact of participation by launching a larger more rigorous study. Investigators have partnered with major organizations providing rehabilitation services for youth as well as key community-based stakeholders including youth, clinicians, and managers, and together investigators plan to further examine whether engaging in an 8-week community-based activity individually chosen by the youth (e.g., sledge hockey, drawing, playing a musical instrument) can lead to a significant improvement in three key body functions: motor, behavioral and emotional. One hundred and fifty youth with physical disabilities living in Quebec and Ontario will participate and engage in an activity of choice. Changes in their body functions (e.g., movement, attention, mood) will be measured multiple times before, during and after engagement in the chosen activity. Findings of this study can guide clinicians, families and policy-makers to select effective approaches that not only promote participation but also facilitate additional motor and mental benefits from a single intervention. Such 'real-world' treatment approaches involving activities of choice can also increase motivation, compliance and reduce burden on the healthcare system and on the youth and families.

DETAILED DESCRIPTION:
Youth with physical disabilities experience restrictions to participation in community-based activities, leading to poor health outcomes. Typical treatment approaches focusing on remediation of impaired body functions ('bottom-up' or upstream approach) have failed to translate into improved participation. As such, reverse 'top-down' participation-based approaches, implemented in one's natural environment, are emerging; yet, their downstream effects have not been established. Specifically, it is unclear whether enhancing participation in self-chosen real-life activity that is meaningful to the youth (e.g., sledge hockey) can simultaneously improve both body functions (e.g., grip strength, attention, anxiety) and activity performance - two key outcomes in pediatric rehabilitation.

Supported by CIHR (2013-17), investigators first proved the effectiveness of PREP intervention (Pathways and Resources for Engagement and Participation) in promoting youth's community participation; then, through SPOR (2017-18) and CIHR Project Grant (2020-23), investigators successfully tested an innovative pragmatic clinical trial to improve body functions through participation. Investigators' promising findings inform the design of this proposed larger more rigorous cross-provincial study called BEYOND, generating sound evidence with widening impact which will serve to support a paradigm shift in clinical practice.

Using PREP, investigators aim to determine the effectiveness of youth engagement in self-chosen 8-week community- based activity program (e.g., drawing, swimming) on change in 3 underlying body functions: motor (using the Functional Reach Test, Trunk Impairment Scale, and dynamometers), behavioral and emotional (using the Behavior Assessment System for Children), and activity performance (via the Canadian Occupational Performance Measure). A 22-week interrupted time series design with multiple baselines across 150 youth with physical disabilities (e.g., cerebral palsy, spina bifida) stratified by sex and severity, aged 12 to 18 living in Quebec and Ontario will be employed. Body functions relevant to each activity will be measured multiple times throughout the entire study and during follow-up, resulting in 450 trajectories of change in body functions (150 youth X 3 functions) and 150 trajectories representing change in activity performance. Mixed-effects models will be used to estimate an intervention effect across youth. Investigators' interdisciplinary team, comprised of researchers in the field of childhood disability and transition-aged youth (occupational therapy, physical therapy, psychology, biostatistics), has partnered with CIUSSS West- Central Montreal and Empowered Kids Ontario, and is well-positioned to accomplish the study objectives.

This novel patient-oriented study will permit drawing firm conclusions to support a shift towards personalized 'top-down' approaches in clinical practice. It will build knowledge that can guide clinicians, families and policy-makers in appraising the benefits of participation-based therapies on improving both functional capacities and performance in meaningful life activities. Demonstrating the multiple benefits generated by one single intervention can facilitate efficient youth-engaging therapies, contributing to the provision of pediatric rehabilitation services. Findings can also enhance knowledge of pragmatic clinical trials for testing complex individual-based interventions that are most appropriate and beneficial for rehabilitation research and practice.

ELIGIBILITY:
Inclusion Criteria:

* a physical disability (e.g., due to cerebral palsy, spina bifida, spinal cord injury, non progressive musculoskeletal disorders, juvenile arthritis);
* restricted mobility, such as an inability to navigate all surfaces and stairs independently and safely without the use of aids, physical assistance, or external support;
* youth with various diagnoses will be eligible;
* youth with cognitive and communication issues and/or intellectual delay will be included and a proxy version of self-reported assessments will be used.
* living in the province of Quebec or Ontario

Exclusion Criteria:

* youth who are recovering within the first year following a severe brain injury or an orthopedic surgery or botulinum toxin treatment 6 months prior or anticipated during the study period
* youth with degenerative disorders
* youth with a severe untreated mental health condition will also be excluded based on the Kessler Psychological Distress Scale (K6)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Behavioral Assessment System for Children | 22 weeks
  Evaluates the behavioral and emotional aspects of body functions using a 4-point scale. T-scores range from 0 to 120 in which lower scores indicate greater behavioral and emotional body functions.
Trunk Impairment Scale | 22 weeks
  Assesses trunk control and includes 3 sub-scales; static sitting balance, dynamic sitting balance and coordination. It contains 17 items rated on a 2-, 3- or 4- point scale. Total score measures motor body functions in terms of trunk control. Total score ranges from 0 (low performance) to 23 (high performance).
Functional Reach Test | 22 weeks
  Assesses motor body functions in terms of reaching. The maximum distance in inches the participant can reach forward while standing/sitting in a fixed position is measured; units: inches.
Jamar/Handheld micro Force Evaluation and Testing 2 (microFET2) Dynamometers | 22 weeks
  Measures motor body functions in terms of maximal grip, pinch strength and isometric muscle strength; units: pounds of force. Scores range from 0 to 200 pounds.
Goniometer | 22 weeks
  Measures active range of motion of specific joints relevant to the activity and based on the task analysis; units: degrees of range of motion.
Canadian Occupational Performance Measure | 22 weeks
  A gold-standard 10-point scale that measures activity performance. Score ranges from 1 (unable to perform) to 10 (performs extremely well).

OTHER OUTCOMES:
Client Satisfaction Questionnaire | This outcome will be assessed once after the intervention (week 22).
  An 8-item tool that measures levels of satisfaction of a program/service using a 4-point scale that takes 3-8 minutes to complete. Overall scores range from 8-32, higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Anaby, PhD, Principal Investigator — McGill University
Locations (1):
- Lethbridge-Layton-Mackay Rehabilitation Center of CIUSSS West-Central Montreal (Mackay site), Montreal, Quebec, Canada